CLINICAL TRIAL: NCT01579422
Title: Social Cognitive Training for Psychosis: Phase I Treatment Development
Brief Title: Social Cognitive Training for Psychosis: Treatment Development
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008007225; 1R34MH090109 (NIH)
Record Dates: First submitted 2012-04-10; First posted 2012-04-18 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia; Psychosis
Keywords: schizophrenia; treatment; social cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- social cognitive training (Experimental)
  Interventions: Behavioral: social cognitive training

INTERVENTIONS:
Behavioral: social cognitive training — social cognitive training, 8-10 sessions

SUMMARY:
The primary aim of this proposal is to develop, refine, manualize and assess the feasibility and preliminary efficacy of a brief, narrowly-focused social cognitive intervention for individuals with psychosis. The intervention will focus on helping individuals interpret social situations, specifically the intentions and feelings of others.

Study methods include preliminary treatment and manual development based on series of uncontrolled cases, manual refinement, and a small feasibility/efficacy trial of the newly developed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or other psychotic disorder
* Age between 18 and 55
* Psychiatrically stable
* Clinician agrees to individual's participation in study
* English as primary language

Exclusion Criteria:

* current (past 30 days) symptoms of alcohol abuse/dependence
* developmental disability
* severe auditory/visual impairment or known neurological disorder
* participant has a legal conservator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
social cognition | change from baseline to approximately 6 weeks
  AIHQ Eyes Task Hinting Task IPSAQ

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States